CLINICAL TRIAL: NCT00762762
Title: The Effect of Periodontal Treatment and the Use of a Triclosan/Copolymer/Fluoride Toothpaste on Glycaemic Control in Diabetics.
Brief Title: Effectiveness of a Triclosan Containing Toothpaste in Maintaining Periodontal Health in a Type 2 Diabetic Population
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2004000685
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2012-04-26 (Estimated); Last update posted 2023-03-03 (Actual); Status verified 2012-04

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Triclosan; hydrated silica gel-based toothpaste; Fluorides

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Total toothpaste (Active Comparator): Brush whole mouth 2x/day for 12 months with triclosan/copolymer/fluoride toothpaste.
  Interventions: Drug: Triclosan/copolymer/fluoride
- Fluoride mouthrinse (Placebo Comparator): Swish whole mouth 2x/day for 12 months with fluoride mouthrinse.
  Interventions: Drug: Fluoride

INTERVENTIONS:
Drug: Triclosan/copolymer/fluoride — Brush whole mouth 2x/day for 12 months with triclosan/copolymer/fluoride toothpaste. Return for required clinical visits @ 12 months for scaling, root planing and donation samples of dental plaque and blood for microbiological analyses.
  Other Names: Total toothpaste
  Arms: Total toothpaste
Drug: Fluoride — Swished around whole mouth twice daily for 12 months. Return for required clinical visits @ 12 months for scaling, root planing and donation samples of dental plaque and blood for microbiological analyses.
  Other Names: Fluorigard oral rinse
  Arms: Fluoride mouthrinse

SUMMARY:
Clinical research study to determine the effectiveness of a triclosan/copolymer/fluoride toothpaste in maintaining periodontal health and therefore glycaemic control in a type 2 diabetic population.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes with poor glycaemic control as evidenced by random blood glucose of >200mg/dl.
* Minimum of 16 teeth
* Chronic periodontitis as indicated by periodontal probing depths >4mm on at least 6 teeth

Exclusion Criteria:

* Any condition requiring antibiotic cover for dental treatment
* Other serious illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Seymour, BDS, PhD, Principal Investigator — Otago University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: all subjects were recruited by the PI at the clinical site.
Pre-assignment Details: all subjects pass a medical exam and meet the study inclusion/exclusion criteria.
Groups:
- Active Comparator: triclosan/fluoride/copolymer toothpaste
- Placebo Comparator: Anti-cavity, fluoride oral rinse
Period: Overall Study
Arm/Group | Active Comparator | Placebo Comparator
Started | 30 | 30
Completed | 24 | 22
Not Completed | 6 | 8
Not completed — Did not return for appointments | 6 | 8

BASELINE CHARACTERISTICS:
Population: Fourteen (14) participants completed baseline data, but did not return for 1 outcome measurement. Lost to follow up.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator | Placebo Comparator | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (7.5) | 48.8 (8.7) | 49.7 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 17 | 17 | 34
Region of Enrollment [Number; unit: participants]
  Australia | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Levels in Blood
Description: Blood is taken from each subject and HbA1c levels were measured at 12 months by Queensland Health Pathology Scientific Services (QHPSS). This test measures the glycated hemoglobin in the blood.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percentage of HbA1c levels in blood
Groups:
- Triclosan/Copolymer/Fluoride Toothpaste: Brush whole mouth 2x/day for 12 months with triclosan/copolymer/fluoride toothpaste.
  Triclosan/copolymer/fluoride: Brush whole mouth 2x/day for 12 months with triclosan/copolymer/fluoride toothpaste. Return for required clinical visits @ 12 months for scaling, root planing and donation samples of dental plaque and blood for microbiological analyses.
Arm/Group | Triclosan/Copolymer/Fluoride Toothpaste | Fluoride Mouthrinse
Number analyzed (Participants) | 30 | 30
percentage of HbA1c levels in blood | 11.42 (1.71) | 10.81 (1.76)
Statistical Analysis 1: Comparison: Triclosan/Copolymer/Fluoride Toothpaste vs Fluoride Mouthrinse; Means and standard deviations. 1 factor ANOVA to balance treatment groups to show no difference between groups. The null hypothesis states that there is no difference between groups; Test type: Other; p = 0.05, ANOVA

2. Primary Outcome: High Sensitivity CRP (C-Reactive Protein)
Description: CRP is a protein found in the blood and is a marker for inflammation in the body. Inflammation plays a role in the initiation and progression of cardiovascular disease.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: µg/ml
Arm/Group | Active Comparator | Placebo Comparator
Number analyzed (Participants) | 30 | 30
µg/ml | 14.94 (13.62) | 10.76 (8.51)
Statistical Analysis 1: Comparison: Active Comparator vs Placebo Comparator; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.05, ANOVA

3. Primary Outcome: C-Peptide
Description: C-Peptide levels in blood indicate whether or not a person is producing insulin
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Active Comparator | Placebo Comparator
Number analyzed (Participants) | 30 | 30
ng/ml | 5.39 (3.68) | 4.61 (0.83)
Statistical Analysis 1: Comparison: Active Comparator vs Placebo Comparator; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.05, ANOVA

4. Primary Outcome: IL-6 (Interleukin - 6)
Description: Levels of Interleukin - 6 (GCF IL-6) found in blood drawn from subjects. Indication of systemic inflammation in the body.(weight in picograms)
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Active Comparator | Placebo Comparator
Number analyzed (Participants) | 30 | 30
pg/ml | 1.93 (1.44) | 2.89 (3.01)
Statistical Analysis 1: Comparison: Active Comparator vs Placebo Comparator; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.05, ANOVA

5. Primary Outcome: TNF-α (Tumor Necrosis Factor - Alpha)
Description: Blood drawn from subjects to determine the level of TNF-α (Tumor necrosis factor - alpha). TNF-α is a pleiotropic inflammatory cytokine involved in systemic inflammation.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Active Comparator | Placebo Comparator
Number analyzed (Participants) | 30 | 30
pg/ml | 4.13 (4.84) | 3.50 (6.41)
Statistical Analysis 1: Comparison: Active Comparator vs Placebo Comparator; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.05, ANOVA

6. Primary Outcome: High Sensitivity CRP (C-Reactive Protein)
Description: as for outcome 2
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: µg/ml
Arm/Group | Active Comparator | Placebo Comparator
Number analyzed (Participants) | 24 | 22
µg/ml | 14.94 (13.62) | 10.76 (8.51)
Statistical Analysis 1: Comparison: Active Comparator vs Placebo Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANOVA

7. Primary Outcome: HbA1c Levels in Blood
Description: as for outcome 1
Time Frame: 12 months
Population: Fourteen (14) participants did not report for 1 year clinical appointment. Lost to follow up.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c levels
Arm/Group | Active Comparator | Placebo Comparator
Number analyzed (Participants) | 24 | 22
percentage of HbA1c levels | 11.42 (1.71) | 10.81 (1.76)
Statistical Analysis 1: Comparison: Active Comparator vs Placebo Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANOVA

8. Primary Outcome: C-Peptide
Description: C-Peptide levels in blood indicate whether or not a person is producing insulin
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Active Comparator | Placebo Comparator
Number analyzed (Participants) | 24 | 22
ng/ml | 5.39 (3.68) | 4.61 (2.70)
Statistical Analysis 1: Comparison: Active Comparator vs Placebo Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANOVA

9. Primary Outcome: IL-6 (Interleukin - 6)
Description: as for outcome 4
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Active Comparator | Placebo Comparator
Number analyzed (Participants) | 24 | 22
pg/ml | 1.93 (1.44) | 2.89 (3.01)
Statistical Analysis 1: Comparison: Active Comparator vs Placebo Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANOVA

10. Primary Outcome: TNF-α (Tumor Necrosis Factor - Alpha)
Description: as for outcome 5
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Active Comparator | Placebo Comparator
Number analyzed (Participants) | 24 | 22
pg/ml | 4.13 (4.84) | 3.50 (6.41)
Statistical Analysis 1: Comparison: Active Comparator vs Placebo Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 12 months (1 years)
Arm/Group | Active Comparator | Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less